CLINICAL TRIAL: NCT01166893
Title: Ability of Modulated Imaging and Laser Speckle Imaging to Determine Burn Wound Severity and Healing Potential
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Anthony Joseph Durkin, Associate Professor, Director, Laboratory for Functional Imaging and Spectroscopy of Superficial Tissues, University of California, Irvine
Other Study IDs: 20097322; R01GM108634 (NIH)
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Skin Burn Multiple
Keywords: burn wound
MeSH Terms: conditions — Burns | interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Burn wound: Modulated Imaging and Laser Speckle Imaging
  Interventions: Device: Modulated Imaging and Laser Speckle Imaging

INTERVENTIONS:
Device: Modulated Imaging and Laser Speckle Imaging — wound healing
  Other Names: MI-LSI developed at UCI Beckman Laser Institute

SUMMARY:
According to the National Burn Repository 2007, the most common type of burn injury is a partial thickness burns. The current standard of care for partial thickness burns is two weeks of topical therapy and wound care. Burns that do not heal within two weeks undergo surgical excision and skin grafting.

DETAILED DESCRIPTION:
Researcher can use the combination of Modulated Imaging and Laser Speckle Imaging can be used as an adjuvant to standard clinical evaluation to gauge burn wound and severity of infection. Researcher can image the burn wounds of and compare with current standard of care, clinical exam, and can use the outcomes information in terms of time to healing and treatment

Modulating Imaging is a noninvasive optical modality measure the metabolic functions of the burn wound.

Laser Speckle Imaging is a noninvasive optical modality can measure blood flow of burn wound.

ELIGIBILITY:
Inclusion Criteria:

1. Male / female all age
2. Subjects is an inpatient or out patient with burn wound

Exclusion Criteria:

1. Subjects cannot lied flat and still for the duration of the imaging
2. Subjects pregnant.

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be selected from University of California Irvine Medical Center Burn Unit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-03; Primary Completion 2028-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Noninvasive burn wound severity assessment | 1 day
  Noninvasive burn wound severity assessment using noncontact optical device

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Durkin, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- UCIMC, Orange, California, United States